CLINICAL TRIAL: NCT02792114
Title: A Phase I Clinical Trial to Evaluate the Safety and Tolerability of Mesothelin-Specific Chimeric Antigen Receptor-Positive T Cells in Patients With Metastatic Mesothelin-Expressing Breast Cancer
Brief Title: T-Cell Therapy for Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-040
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Metastatic HER2-negative Breast
Keywords: T-Cell; Chimeric antigen receptor (CAR); CAR T cells; Triple-negative breast cancer; Immunotherapy T-cell therapy; 16-040; immunotherapy; CAR
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Cyclophosphamide; AP 1903 reagent

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T-cell infusion (Experimental): A single blood volume leukapheresis for harvesting of PBMCs will be performed, As the transduced T cells will be frozen, the timing of leukapheresis is not defined & can vary from patient to patient. Subsequently, a single dose of mesothelin-targeted T cells will be infused via intravenous catheter or central line (i.e., mediport). Patients will be monitored in the hospital and discharged home after a minimum of 48 hours. Patients will be monitored closely as outpatients for the next 2 months. Patients will be followed weekly as outpatients for the first 8 weeks after treatment. All patients will be hydrated intravenously, premedicated with acetaminophen & diphenhydramine, & administered cyclophosphamide at 1.5 g/m2 2 to 7 days (Day -7 to Day -2) before administration of mesothelin-targeted T cells.
  Interventions: Drug: Cyclophosphamide; Biological: Mesothelin-targeted T cells; Drug: AP1903

INTERVENTIONS:
Drug: Cyclophosphamide
Biological: Mesothelin-targeted T cells
Drug: AP1903

SUMMARY:
The purpose of this study is to test the safety of different doses of specially prepared T cells collected from the blood. The investigators want to find a safe dose of these modified T cells for patients who have metastatic HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with metastatic breast cancer
* Karnofsky performance status ≥70%
* Patients with breast cancer that is pathologically confirmed at MSKCC (pathology from outside institutions is acceptable for the screening phase of the protocol) and defined by the following:

  * HER2 negative (in cases of mixed HER2 results, the most recent pathology results considered reflective of the active cancer will be considered)
  * Previously treated with at least 1 chemotherapy regimen for metastatic disease and documented progression
* Expression of mesothelin must be confirmed by meeting 1 of the following criteria:

  * Mesothelin expression (>10% of the tumor expressing mesothelin) by IHC
  * Elevated serum SMRP levels (>1.0 nM/L)
* Presence of measurable or evaluable disease
* Chemotherapy, targeted therapy (such as a tyrosine kinase inhibitor), or radiotherapy must have been completed at least 14 days before administration of T-cells. Prior immunotherapy with checkpoint blockade (i.e., PD1 inhibitor, PDL1 inhibitor, or CTL4-antagonist or similar agent) must have been completed more than 1 month before the T-cell infusion.

  *Chemotherapy must have been completed at least 7 days prior to leukapheresis
* Any major operation must have occurred at least 28 days before study enrollment.
* All acute toxic effects of any previous radiotherapy, chemotherapy, or surgical procedures must have resolved to grade 1 or lower according to CTCAE
* Lab requirements (hematology):

  * White blood cell (WBC) count ≥3000 cells/mm^3
  * Absolute neutrophil count ≥1500 neutrophils/mm^3
  * Platelet count ≥100,000 platelets/mm^3
* Lab requirements (serum chemistry):

  * Bilirubin <1.5x upper limit of normal (ULN)
  * Serum alanine aminotransferase/serum aspartate aminotransferase (ALT/AST) <5x ULN
  * Serum creatinine <1.5x ULN or Cr >1.5x ULN, but calculated clearances of >60
* Negative screen for human immunodeficiency virus (HIV), hepatitis B virus (HBV) antigen, and hepatitis C virus (HCV). If testing was performed during the previous 3 months, there is no need to repeat testing, as long as documentation of results is provided to the study site. Subjects must receive counseling and sign a separate informed consent form for HIV testing.
* Subjects and their partners with reproductive potential must agree to use an effective form of contraception during the period of drug administration and for 4 weeks after completion of the last administration of the study drug. An effective form of contraception is defined as oral contraceptives plus 1 form of barrier or double-barrier method contraception (condom with spermicide or condom with diaphragm).
* Subjects must be able to understand the potential risks and benefits of the study and must be able to read and provide written, informed consent for the study.
* Availability of archival tumor tissues (FFPE tissue block or 10-15 unstained slides)

Exclusion Criteria:

* Untreated or active CNS metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control); patients with a history of treated CNS metastases are eligible, provided that all of the following criteria are met:

  * Presence of measurable or evaluable disease outside of the CNS;
  * Radiographic demonstration of improvement upon completion of CNS- directed therapy and no evidence of interim progression between completion of CNS-directed therapy and the screening radiographic study;
  * Completion of radiotherapy ≥8 weeks prior to the screening radiographic study;
  * Discontinuation of corticosteroids and anticonvulsants ≥4 weeks prior to the screening radiographic study.
* History of seizure disorder
* Patients currently receiving treatment for concurrent active malignancy. Prior immunotherapy with checkpoint blockade (i.e., PD1 inhibitor, PDL1 inhibitor, or CTL4-antagonist or similar agent) must have been completed more than 1 month prior to the T-cell infusion.
* Autoimmune or antibody-mediated disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, ulcerative colitis, Crohn's disease, and temporal arteritis (patients with a history of hypothyroidism will not be excluded)
* Clinically significant cardiac disease (New York Heart Association class III/IV) or severe debilitating pulmonary disease
* Pregnant or lactating women
* Known active infection requiring antibiotics within 7 days of the start of treatment (Day 0)
* A requirement for daily systemic corticosteroids for any reason or a requirement for other immunosuppressive or immunomodulatory agents. Topical, nasal, and inhaled steroids are permitted.
* Administration of live, attenuated vaccine within 8 weeks before the start of treatment (Day 0) and throughout the study
* Any other medical condition that, in the opinion of the PI, may interfere with a subject's participation in or compliance with the study
* Participation in a therapeutic research study or receipt of an investigational drug within 30 days of T-cell infusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated does (MTD) | 2 years
  We have designed the dose-escalation using a standard 3+3 design. In this design, patients will be treated in sequential groups of 3 to 6 patients per T cell dose. With 4 dose levels, the projected trial size for this study is a minimum of 4 and a maximum of 24 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shanu Modi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center (Consent and follow-up only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and follow-up only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and follow-up only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack (Consent and follow-up only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and follow-up only), East White Plains, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-Up only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/